CLINICAL TRIAL: NCT05994157
Title: Phase 1, Open-label, Dose-escalation Trial with CD38-SADA:177 Lu-DOTA Drug Complex in Subjects with Relapsed or Refractory Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Y-mAbs Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1201
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Non-hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CD38-SADA:177Lu-DOTA Complex (Experimental)
  Interventions: Drug: CD38-SADA:177Lu-DOTA Complex

INTERVENTIONS:
Drug: CD38-SADA:177Lu-DOTA Complex — The IMP is a two-step radioimmunotherapy, delivered as two separate products CD38-SADA and 177Lu-DOTA. Both will be administered as an IV infusions.

SUMMARY:
Patients with non-Hodgkin Lymphoma will be treated with CD38-SADA:177Lu-DOTA complex (The IMP is a two-step radioimmunotherapy, delivered as two separate products CD38-SADA and 177Lu-DOTA) to establish optimal and safe therapeutic doses and dosing schedule of CD38-SADA, and 177Lu-DOTA.

ELIGIBILITY:
Inclusion Criteria:

* Target population must have relapsed, progressive or refractory non-hodgkin lymphoma and be ineligible for or have exhausted standard therapeutic options that may prolong survival
* The subject must have fluoro-deoxyglucose (FDG)-avid lymphoma with measurable disease
* CD38 positive tumor at most recent biopsy (new or archival) documented at central laboratory
* Subject must have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
* Each subject must sign an ICF indicating that he or she understands the purpose of, and procedures required for the trial and is willing to participate in the trial.

Exclusion Criteria:

* Primary central nervous system lymphoma or known central nervous system involvement with lymphoma
* Systemic chemotherapy, radiotherapy, immunotherapy, or major surgery administered within 3 weeks (for nitrosoureas within 6 weeks) prior to the first dose of CD38-SADA
* Radioimmunotherapy within 100 days prior to the first dose of CD38-SADA
* Autologous stem cell transplantation within 42 days prior to the first dose of CD38-SADA
* Treatment with approved CAR-T within 100 days prior to the first dose of CD38-SADA
* >40% lymphoma bone marrow involvement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Tumor imaging and occurrence of dose limiting toxicities (DLT) during the DLT evaluation period (Part A) | 4 weeks
Occurrence of dose limiting toxicities during the DLT evaluation period (Part B) | 4 weeks

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - HonorHealth, Scottsdale, Arizona
  - City of Hope, Duarte, California
  - Corewell Health-BAMF Health, Grand Rapids, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Stony Brook Cancer Center, Stony Brook, New York
  - East Carolina University Leo W. Jenkins Cancer Center, Greenville, North Carolina

IPD SHARING:
Plan to Share IPD: No